CLINICAL TRIAL: NCT04193696
Title: Combining Radiation Therapy With Anti-PD-1 for Patients With Advanced Hepatocellular Carcinoma (RT+PD-1-HCC)
Brief Title: RT+ Anti-PD-1 for Patients With Advanced HCC (RT+PD-1-HCC)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Jian-Hong Zhong, Professor, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RT+PD-1-HCC
Record Dates: First submitted 2019-12-09; First posted 2019-12-10 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Hepatocellular Carcinoma
Keywords: advanced HCC; anti-PD-1; radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: This stuy has only one arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy plus PD-1 (Experimental)
  Interventions: Drug: Radiation therapy and systemic anti-PD-1 immunotherapy for patients with advanced hepatocellular carcinoma

INTERVENTIONS:
Drug: Radiation therapy and systemic anti-PD-1 immunotherapy for patients with advanced hepatocellular carcinoma — The treatment will be started within 1 week after being admitted into the trial. IMRT or SBRT are adopted , and dose of radiation: Dt-PGTV=40Gy/10fractions,Dt-PGTV=30Gy/10fractions,Dt-PGTV=20Gy/10fractions ,and so on.200mg/ of Carelizumab for injection will be given intravenously every 3 weeks for 5 times since the first day of radiotherapy until disease progression, or intolerable toxicity.

SUMMARY:
Hepatocellular carcinoma (HCC) is a common malignancy, and its incidence is expected to increase in many countries in coming decades. Approximately 70-80% of newly diagnosed HCC patients already have advanced disease. Sorafenib and lenvatinib are recommended as first-line options for advanced HCC, the median overall survival of the patients with advanced HCC receiving sorafenib reached 10.7 months. Based on the results of phase II clinical studies and the recommendation of guidelines, the PD-1 monoclonal antibody, such as nivolumab and pembrolizumab, have been approved to treat the patients with advanced HCC by the FDA. PD-1 monoclonal antibody has been recommended as a second-line therapeutic strategy for HCC in the 2018 CSCO guidelines for the diagnosis and treatment of primary liver cancer. However, the results of existing studies indicate that the objective response rate (ORR) of first-line PD-1 antibody therapy for patients with advanced liver cancer is about 20%.

There is a growing recognition of radiation-induced cancer cells-external tumor control mechanisms, in which radiation therapy(RT) contributes not only to local control of target lesions, but also to the control of metastases away from the treatment site. In recent years, RT combined with immunotherapy as a new treatment method has achieved certain curative effect in some patients with metastatic cancer. Therefore, it is interesting to investigate the efficacy of combining radiation therapy plus systemic anti-PD-1 immunotherapy for patients with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Diagnosis of advanced HCC was confirmed by histopathological examination or clinical diagnosis, consistent with the following two conditions:

  1. Extrahepatic metastasis with more than one measurable lesion;
  2. Intrahepatic multifocal lesions with more than one measurable lesion independent of the radiosurgery field
* Patients have Child-Pugh A liver function
* Expected survival ≥ 3 months
* Unwilling to receive or unable to tolerate first-line treatment with sorafenib

Exclusion Criteria:

* History of other malignancy
* History of systemic immunotherapy
* History of Radiation therapy within 6 months before the first administration
* History of active autoimmune diseases requiring systemic treatment within 2 years before recruiting.
* There are active infections that require systemic treatment
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients
* Diagnosed with immunodeficiency or receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days before the first administration of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-01-10 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-07-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 6 months

SECONDARY OUTCOMES:
Overall survival | 1 year
Abscopal effects rate | 6 months

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Background] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Background] Zhu AX, Finn RS, Edeline J, Cattan S, Ogasawara S, Palmer D, Verslype C, Zagonel V, Fartoux L, Vogel A, Sarker D, Verset G, Chan SL, Knox J, Daniele B, Webber AL, Ebbinghaus SW, Ma J, Siegel AB, Cheng AL, Kudo M; KEYNOTE-224 investigators. Pembrolizumab in patients with advanced hepatocellular carcinoma previously treated with sorafenib (KEYNOTE-224): a non-randomised, open-label phase 2 trial. Lancet Oncol. 2018 Jul;19(7):940-952. doi: 10.1016/S1470-2045(18)30351-6. Epub 2018 Jun 3. PMID 29875066
- [Background] El-Khoueiry AB, Sangro B, Yau T, Crocenzi TS, Kudo M, Hsu C, Kim TY, Choo SP, Trojan J, Welling TH Rd, Meyer T, Kang YK, Yeo W, Chopra A, Anderson J, Dela Cruz C, Lang L, Neely J, Tang H, Dastani HB, Melero I. Nivolumab in patients with advanced hepatocellular carcinoma (CheckMate 040): an open-label, non-comparative, phase 1/2 dose escalation and expansion trial. Lancet. 2017 Jun 24;389(10088):2492-2502. doi: 10.1016/S0140-6736(17)31046-2. Epub 2017 Apr 20. PMID 28434648
- [Background] Herrera FG, Bourhis J, Coukos G. Radiotherapy combination opportunities leveraging immunity for the next oncology practice. CA Cancer J Clin. 2017 Jan;67(1):65-85. doi: 10.3322/caac.21358. Epub 2016 Aug 29. PMID 27570942
- [Background] Twyman-Saint Victor C, Rech AJ, Maity A, Rengan R, Pauken KE, Stelekati E, Benci JL, Xu B, Dada H, Odorizzi PM, Herati RS, Mansfield KD, Patsch D, Amaravadi RK, Schuchter LM, Ishwaran H, Mick R, Pryma DA, Xu X, Feldman MD, Gangadhar TC, Hahn SM, Wherry EJ, Vonderheide RH, Minn AJ. Radiation and dual checkpoint blockade activate non-redundant immune mechanisms in cancer. Nature. 2015 Apr 16;520(7547):373-7. doi: 10.1038/nature14292. Epub 2015 Mar 9. PMID 25754329
- [Derived] Li JX, Su TS, Gong WF, Zhong JH, Yan LY, Zhang J, Li LQ, He ML, Zhang RJ, Du YQ, Wang XT, Liang SX, Xiang BD. Combining stereotactic body radiotherapy with camrelizumab for unresectable hepatocellular carcinoma: a single-arm trial. Hepatol Int. 2022 Oct;16(5):1179-1187. doi: 10.1007/s12072-022-10396-7. Epub 2022 Aug 24. PMID 36001228